CLINICAL TRIAL: NCT06373107
Title: Investigating Effects of High-intensity Gait Training on Gait Function, Balance and Depression Following Stroke and the Impact of Social Determinants of Health and Depression on Patients' Adherence to Physical Therapy
Brief Title: Investigating Effects of High-intensity Gait Training on Gait, Balance and Depression Post-stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participants
Sponsor: Alvernia University (Other)
Collaborators: Lehigh Valley Health Network (Other)
Responsible Party: Principal Investigator, Soo Yeon Sun, PT, PhD, Associate Professor, Alvernia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2117651-2
Record Dates: First submitted 2024-03-25; First posted 2024-04-18 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: High intensity gait training; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High intensity gait training (Experimental): Participants will receive 20 sessions of vigorous walking practice. These sessions are 2-3 times a week.
  Interventions: Behavioral: High intensity gait training

INTERVENTIONS:
Behavioral: High intensity gait training — Participants will practice walking that is vigorous enough to keep their heart rate over a certain level during their physical therapy sessions. During the sessions, participants will walk and step vigorously enough to keep the heart rate between 60-80% of their maximum heart rate. Maintaining this heart rate during exercise helps to improve heart health and walking, which can affect people after a stroke.

SUMMARY:
The purpose of this research is to study the improvements from walking practice that is vigorous enough to keep participants' heart rate over a certain target level during their physical therapy sessions. The investigators want to know about improvements in participants' walking function and mental health after 20 interventions. The study also aims to evaluate if participants' mental health, social support, and health literacy affect their attendance at physical therapy sessions.

DETAILED DESCRIPTION:
The purpose of this research is to study the improvements from walking practice that is vigorous enough to keep participants' heart rate over a certain target level during their physical therapy sessions. The investigators want to know about improvement in participants' walking function and mental health after 20 interventions. The study also aims to evaluate if participants' mental health, social support, and health literacy affect their attendance at physical therapy sessions.

The findings from this study will help the researchers and clinicians decide how to help people with stroke better. Further, the findings will determine how depressive symptoms, health literacy, and other factors such as language and education affect attendance to therapy.

About 24 subjects will take part in this research.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English or Spanish speaking
* A diagnosis of stroke (intracerebral hemorrhage or acute ischemic stroke)
* Referred to LVHN Outpatient Neurologic Rehab (hereafter referred to as outpatient PT)

Exclusion Criteria:

* Unable to follow 1-step commands
* > 220 pounds (100 kg)
* Height < 5'0" or > 6'4"
* Unable to take a few steps with assistance
* A score of ≥ 50/56 on Berg Balance Scale (BBS)
* A score of ≥ 26/30 on Functional Gait Assessment (FGA)
* Resting blood pressure >180/110 mmHg
* Resting heart rate > 120 bpm
* Severe cardiac disease (New York Heart Association Classification IV)
* Severe spasticity (Modified Ashworth score > 3)
* Unstable spine or unhealed pelvic/limb fractures
* Active heterotrophic ossification impacting lower extremity range of motion
* Significant lower or upper extremity contractures
* Inability to achieve neutral ankle dorsiflexion with 12° of knee flexion
* Pregnancy
* Colostomy
* Poor skin integrity
* Unresolved deep vein thrombosis
* Lower limb prosthesis or amputation
* Leg length discrepancies > 0.5 inches for upper legs, 0.75 inches for lower legs
* ROM restrictions preventing normal, reciprocal gait
* Inability to stand for > 3 minutes due to pain or orthostatic hypotension
* Pusher syndrome
* Cortical blindness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
3-meter backwards walk test | Pre-, mid- (week 5) and post-intervention (within 2 weeks after the conclusion of intervention)
  Measures backward gait velocity
6-minute walk test | Pre-, mid- (week 5) and post-intervention (within 2 weeks after the conclusion of intervention)
  Measures aerobic capacity and endurance
10-meter walk test | Pre-, mid- (week 5) and post-intervention (within 2 weeks after the conclusion of intervention)
  Measures forward gait velocity
Surface electromyography (EMG) | Pre-, mid- (week 5) and post-intervention (within 2 weeks after the conclusion of intervention)
  Electromyographical recording of 8 leg muscles () is done during forward and backward walking tests.The EMG will be recorded during 3-meter Backward Walk Test, 6-minute Walk Test, and 10-meter Walk Test in all participants
Berg Balance Scale | Pre-, mid- (week 5) and post-intervention (within 2 weeks after the conclusion of intervention)
  a 14-item objective measure that assesses static balance and fall risk in adults. Berg balance scale scoring ranges from 0 to 56, with higher scores mean a better outcome.
Functional Gait Assessment | Pre-, mid- (week 5) and post-intervention (within 2 weeks after the conclusion of intervention)
  This scale assess postural stability during walking and assesses an individual's ability to perform multiple motor tasks while walking. Scoring for each FGA item ranges from 0 for severe impairment to 3 for normal performance. The highest score possible is 30, with higher scores correlating better gait function.
Borg Rating Scale of Perceived Exertion (RPE) | Pre-, mid- (week 5) and post-intervention (within 2 weeks after the conclusion of intervention)
  RPE is used to prescribe and monitor exercise intensity and correlates well with physiological measures of exercise intensity, including heart rate. The Borg Rating Scale of Perceived Exertion will be measured in all participants at the completion of 6 Minute Walk test. It ranges from 6 to 20, where 6 means "no exertion at all" and 20 means "maximal exertion." A lower score indicates a better exercise endurance.
Patient Health Questionnaire (PHQ-9) | Pre-, mid- (week 5) and post-intervention (within 2 weeks after the conclusion of intervention)
  Depressive symptom questionnaire. As a severity measure, the PHQ-9 score can range from 0 to 27, since each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day). A lower score indicates less depressive symptoms.
Rate of patient attendance (Compliance) to physical therapy | Participant's attendance to physical therapy is tracked throughout the intervention sessions.
  Greater than or equal to 80% attendance to physical therapy is considered compliance to physical therapy.
Newest Vital Sign | Pre-intervention (baseline)
  The NVS is a 6-question screening tool that identifies participants' risk of low or limited health literacy based on interpreting an ice cream nutrition label. It is available from Pfizer Pharmaceutical Company. The level of health literacy for each individual will be categorized based on the scores: a score of 0-1 suggests a high likelihood of limited literacy, a score of 2-3 indicates the possibility of limited literacy, and a score of 4-6 almost always indicates adequate literacy. This categorical variable will be used to determine the association with adherence to physical therapy.
Multidimensional Scale of Perceived Social Support (MSPSS) | Pre-intervention (baseline)
  The MSPSS is a 12-item self-administered scale that measures social support. It contains 12-items, rated on a 7-point Likert-type scale, ranging from 1 "very strongly disagree" to 7 "very strongly agree." The scale was divided into 3 subscales: family, friends, and significant other, with each section consisting of 4 items. The response scale ranges from 12 to 84. Higher scores indicate a greater family social support.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Yeon Sun, PhD, Principal Investigator — Alvernia University
Locations (1):
- Lehigh Valley Health Network Outpatient Neurologic Rehab, Allentown, Pennsylvania, United States